CLINICAL TRIAL: NCT02616952
Title: Effect of Yiqi Suoquan Tang, a Chinese Herbal Decoction, on Stress Urinary Incontinence
Brief Title: A Chinese Herbal Decoction for Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ran Pang, Associate Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014S292
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Urinary Incontinence, Stress
Keywords: Stress urinary incontinence; Chinese Herb; Traditional Chinese medicine; Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chinese herbal therapy group (Experimental): Participants take a Chinese herbal decoction, Yiqi Suoquan Tang, 200ml orally twice a day for 12 weeks.
  Interventions: Dietary Supplement: Chinese herbal therapy
- Pelvic floor muscle training group (Other): Pelvic floor muscle training includes intensive exercises and home exercises. Intensive exercises are conducted in hospital once a week while home exercises are performed three times daily for 12 weeks.
  Interventions: Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Dietary Supplement: Chinese herbal therapy — Participants take a Chinese herbal decoction, Yiqi Suoquan Tang, 200ml orally twice a day for 12 weeks. The Yiqi Suoquan Tang are composed of Radix Astragali 30 g, Radix Codonopsis pilosula 10g, Radix Angelica sinensis 10g, Radix Atractylodis Macrocephalae 10g, Fructus Alpiniae Oxyphyllae 10g, Radix Lindera aggregata 6g, Rhizoma Dioscoreae 10g, pericarpium citri reticulatae 10g, Rhizoma Cimicifuga 10g, Radix Bupleuri 10g, Fructus Rubi 15g, and Semen raphani 10g. All the decoctions are provided by the Department of Pharmacy, Guang'anmen Hospital, China Academy of Chinese Medical Sciences, and are packed in opaque plastic bags with 200 ml for each one.
  Other Names: Yiqi Suoquan Tang
  Arms: Chinese herbal therapy group
Behavioral: Pelvic floor muscle training — In intensive exercises, participants are taught how to identify the muscles: 1) identify anal sphincter/feel anus, and try to raise it from chair (without adding abdominal, thigh, and buttock muscles) with a position of sitting; 2) identify levator ani and try to raise vagina from chair (without adding abdominal, thigh, and buttock muscles) with a position of Sitting, bent forward, elbows on knees; 3) contract levator ani with a position of sitting, lying, and standing; 4) contract anal sphincter with a position of sitting, lying, and standing. Once the participants can identify the muscles, they are asked to do a set consists of 10 contractions, each lasting 5 seconds, with a 5 seconds break between contractions. Then they need to do same procedure 3 times daily as the home exercises.
  Other Names: Kegel Exercise
  Arms: Pelvic floor muscle training group

SUMMARY:
The purpose of this study is to determine whether Yiqi Suoquan Tang, a Chinese Herbal decoction, is effective in the treatment of female stress urinary incontinence.

DETAILED DESCRIPTION:
The pilot randomized, controlled trial is aimed to preliminarily assess the effectiveness of Yiqi Suoquan Tang, a Chinese Herbal decoction, in the treatment of female stress urinary incontinence (SUI). Eligible participants will be randomly allocated to receiving Yiqi Suoquan Tang or pelvic floor muscle training (PFMT) using a random number generator in a 1:1 ratio. To minimize the evaluation bias, the outcome assessors and statisticians will be masked to treatment allocation.

Assuming a two-sided alpha of 0.05, power of 90%, and a 20% drop-out, a sample size of 36 would be needed for each group. The statistical analysis will be performed based on the intention-to-treat principle, which is defined as patients that have received at least one treatment. Missing data will be replaced by the last observed value. Continuous variables will be compared by Student t test or Mann-Whitney U test; categorical variables will be analyzed by chi-square test, Fisher's exact test or Kruskal-Wallis H test as appropriate. For comparison between two time points, paired t-test or Wilcoxon signed rank test will be used as appropriate. A statistically significant difference was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stress urinary incontinence
* Must be able to swallow Chinese hebal decoction

Exclusion Criteria:

* Urinary tract infection
* Neurogenic bladder
* Pelvic organ prolapse > stage 2
* Overactive bladder
* Previous anti-incontinence surgery
* Post-void residual urine volume (PVR) > 100ml.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in 24h pad testing | 12 weeks

SECONDARY OUTCOMES:
Change in ICIQ-SF questionnaire | 12 weeks
Change in abdominal leak-point pressure | 12 weeks
Change in I-QOL questionnaire | 12 weeks

OTHER OUTCOMES:
Adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ran Pang, MD, Principal Investigator — Guang'anmen hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China